CLINICAL TRIAL: NCT03781596
Title: Randomized Controlled Trial Comparing Fluticasone Plus Omeprazole With Fluticasone Alone for Eosinophilic Esophagitis
Brief Title: EoE RCT Fluticasone and Omeprazole vs Fluticasone Alone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Claire Daniels (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Claire Daniels, Associate Investigator, Walter Reed National Military Medical Center
Organization: Walter Reed National Military Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: WRNMMC-2018-0133
Record Dates: First submitted 2018-11-11; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Fluticasone; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluticasone and omeprazole (Experimental): These patients will be prescribed swallowed fluticasone and omeprazole to be taken together for the 8 week period. Dosing will be based on weight and age. Primary outcome measure will be the change in esophageal biopsy histology, or number of eosinophils per high powered field, from week 0 to week 8. Secondary outcomes will include changes in the following variables between week 0 and 8: eotaxin staining of the esophageal biopsy tissue, endoscopic scoring from photos of the esophagus obtained during endoscopy, and symptom scoring based on surveys.
  Interventions: Diagnostic Test: Retrospective evaluation of endoscopy prior to study drug; Other: Symptom Survey; Other: Medication Compliance Phone Call; Diagnostic Test: Endoscopy while on study drug; Drug: Fluticasone; Drug: Omeprazole
- Fluticasone and placebo (Placebo Comparator): These patients will be prescribed swallowed fluticasone and a placebo medication that appears identical to omeprazole to be taken together for an 8 week period. Dosing will be based on weight and age. Primary outcome measure will be the change in esophageal biopsy histology, or number of eosinophils per high powered field, from week 0 to week 8. Secondary outcomes will include changes in the following variables between week 0 and 8: eotaxin staining of the esophageal biopsy tissue, endoscopic scoring from photos of the esophagus obtained during endoscopy, and symptom scoring based on surveys.
  Interventions: Diagnostic Test: Retrospective evaluation of endoscopy prior to study drug; Other: Symptom Survey; Other: Medication Compliance Phone Call; Diagnostic Test: Endoscopy while on study drug; Drug: Fluticasone; Drug: Placebo oral capsule

INTERVENTIONS:
Diagnostic Test: Retrospective evaluation of endoscopy prior to study drug — Once enrolled, the patient's original endoscopy will be evaluated including the images from the EGD and the biopsies for eotaxin 3 staining and eosinophilic burden.
Other: Symptom Survey — Patient will complete symptom survey prior to starting the study drugs.
Other: Medication Compliance Phone Call — The patient will receive a phone call at 4 weeks to evaluate medication compliance including the number on the inhaler and the number of pills remaining in the container.
Diagnostic Test: Endoscopy while on study drug — Endoscopy will be performed after 8 weeks of therapy. Endoscopic scoring will be assigned and the histology will be evaluated, including eotaxin 3 staining. The change in eosinophil count and eotaxin staining will be measured.
Other: Symptom Survey — The patient will complete a symptom survey after 8 weeks on the study drugs, and the change in survey score will be measured.
Drug: Fluticasone — Participants in the experimental and placebo arms will be given swallowed fluticasone for an 8 week course. Doses determined by age and weight.
Drug: Omeprazole — The participants in the experimental arm will be given oral omprazole capsules for an 8 week period (along with the swallowed fluticasone). Doses determined by age and weight.
  Arms: Fluticasone and omeprazole
Drug: Placebo oral capsule — The participants in the placebo arm will be given placebo capsules for an 8 week period (along with the swallowed fluticasone). Number of pills determined by age and weight (to match omeprazole dosing).
  Arms: Fluticasone and placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of combination therapy with omeprazole and swallowed fluticasone vs fluticasone therapy and placebo in the treatment of Eosinophilic Esophagitis (EoE) in children and adults. This study will be a double-blinded, randomized controlled trial. The primary outcome measured will be histologic assessment of esophageal tissue biopsies measuring number of eosinophils per high power field (eos/hpf). Secondary outcomes will be endoscopic findings and symptomatic changes following therapy using validated endoscopic scoring measures and participant surveys, respectively.

DETAILED DESCRIPTION:
Subjects that meet study inclusion criteria will be recruited from the Adult and Pediatric Gastroenterology clinics at Walter Reed National Military Medical Center through routine clinic visits, will meet with an investigator, and complete informed consent/assent. The participants will then complete a validated clinical symptom reporting tool - the Eosinophilic Esophagitis symptom activity index (EEsAI) for age 18 and above, or the Pediatric Quality of Life Inventory (PedsQL) for age 6-17yrs - and have their initial Esophagogastroduodenoscopy (EGD) images evaluated via a validated Endoscopic Reference Score (EREFS). Esophageal biopsies taken at the patient's initial EGD will be assessed by 2 designated blinded pathologists to record the number of eosinophils per high power field (HPF), as well as perform tissue immunohistochemical staining for eotaxin-3. Participants will be block randomized to treatment or control groups and complete 8 weeks of therapy, with a phone follow up at 4 weeks for medication compliance. At the completion of 8 weeks of therapy, the participants will have repeat EGD to assess for mucosal healing, which is the standard of care in the treatment of EoE. At this EGD, the images will be assigned an EREFS and the biopsies will be evaluated for eosinophils per high powered field and eotaxin-3 staining. The patient will also complete an EEsAI or PedsQL. This procedure will end the 8 week study period.

ELIGIBILITY:
Inclusion Criteria:

* age 6 to 60 years old
* DEERS (defense enrollment eligibility reporting system) eligible
* diagnosis of eosinophilic esophagitis

Exclusion Criteria:

* Outside of age range
* Co-existing inflammatory gastroenterologic condition such as celiac disease, eosinophilic esophagitis, or inflammatory bowel disease.
* Concurrent use of oral steroids
* Pregnancy
* Refusal to undergo endoscopy

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-10-02 (Estimated); Study Completion 2022-10-02 (Estimated)

PRIMARY OUTCOMES:
Change in esophageal eosinophilia | There will be one at week 0 and week 8.
  The number of eosinophils per high powered field will be counted by participating pathologist.

SECONDARY OUTCOMES:
Change in Endoscopic Reference Score | This will be done at week 0 and week 8
  Endoscopic appearance will be evaluated with a validated scoring method: Minimum score 0, maximum score 10. Scores come from 5 outcomes: Fixed rings (0-3 points), exudates (0-2 points), furrows (0-2 points), edema (0-2 points), stricture (0-1 points).
Change in Symptom Scoring | Week 0 and week 8
  Clinical changes will be evaluated by either one of 2 validated tools: Eosinophilic Esophagitis symptom activity index (EEsAI) for age 18 and above, or the Pediatric Quality of Life Inventory (PedsQL) for age 6-17yrs.
  Both of these tools are considered proprietary and we have permission from the companies to use this scoring system for research - and their grading scales were provided. Copyright for PedsQL - JW Varni 1998. Confidentiality for EEsAI scoring - EEsAI Study Group at the University of Bern.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liacouras CA, Furuta GT, Hirano I, Atkins D, Attwood SE, Bonis PA, Burks AW, Chehade M, Collins MH, Dellon ES, Dohil R, Falk GW, Gonsalves N, Gupta SK, Katzka DA, Lucendo AJ, Markowitz JE, Noel RJ, Odze RD, Putnam PE, Richter JE, Romero Y, Ruchelli E, Sampson HA, Schoepfer A, Shaheen NJ, Sicherer SH, Spechler S, Spergel JM, Straumann A, Wershil BK, Rothenberg ME, Aceves SS. Eosinophilic esophagitis: updated consensus recommendations for children and adults. J Allergy Clin Immunol. 2011 Jul;128(1):3-20.e6; quiz 21-2. doi: 10.1016/j.jaci.2011.02.040. Epub 2011 Apr 7. PMID 21477849
- [Background] Dellon ES, Jensen ET, Martin CF, Shaheen NJ, Kappelman MD. Prevalence of eosinophilic esophagitis in the United States. Clin Gastroenterol Hepatol. 2014 Apr;12(4):589-96.e1. doi: 10.1016/j.cgh.2013.09.008. Epub 2013 Sep 11. PMID 24035773
- [Background] Liacouras CA, Wenner WJ, Brown K, Ruchelli E. Primary eosinophilic esophagitis in children: successful treatment with oral corticosteroids. J Pediatr Gastroenterol Nutr. 1998 Apr;26(4):380-5. doi: 10.1097/00005176-199804000-00004. PMID 9552132
- [Background] Schaefer ET, Fitzgerald JF, Molleston JP, Croffie JM, Pfefferkorn MD, Corkins MR, Lim JD, Steiner SJ, Gupta SK. Comparison of oral prednisone and topical fluticasone in the treatment of eosinophilic esophagitis: a randomized trial in children. Clin Gastroenterol Hepatol. 2008 Feb;6(2):165-73. doi: 10.1016/j.cgh.2007.11.008. PMID 18237866
- [Background] Papadopoulou A, Dias JA. Eosinophilic esophagitis: an emerging disease in childhood - review of diagnostic and management strategies. Front Pediatr. 2014 Nov 21;2:129. doi: 10.3389/fped.2014.00129. eCollection 2014. PMID 25485261
- [Background] Konikoff MR, Noel RJ, Blanchard C, Kirby C, Jameson SC, Buckmeier BK, Akers R, Cohen MB, Collins MH, Assa'ad AH, Aceves SS, Putnam PE, Rothenberg ME. A randomized, double-blind, placebo-controlled trial of fluticasone propionate for pediatric eosinophilic esophagitis. Gastroenterology. 2006 Nov;131(5):1381-91. doi: 10.1053/j.gastro.2006.08.033. Epub 2006 Aug 16. PMID 17101314
- [Background] Dohil R, Newbury R, Fox L, Bastian J, Aceves S. Oral viscous budesonide is effective in children with eosinophilic esophagitis in a randomized, placebo-controlled trial. Gastroenterology. 2010 Aug;139(2):418-29. doi: 10.1053/j.gastro.2010.05.001. Epub 2010 May 7. PMID 20457157
- [Background] Butz BK, Wen T, Gleich GJ, Furuta GT, Spergel J, King E, Kramer RE, Collins MH, Stucke E, Mangeot C, Jackson WD, O'Gorman M, Abonia JP, Pentiuk S, Putnam PE, Rothenberg ME. Efficacy, dose reduction, and resistance to high-dose fluticasone in patients with eosinophilic esophagitis. Gastroenterology. 2014 Aug;147(2):324-33.e5. doi: 10.1053/j.gastro.2014.04.019. Epub 2014 Apr 22. PMID 24768678
- [Background] Alexander JA, Jung KW, Arora AS, Enders F, Katzka DA, Kephardt GM, Kita H, Kryzer LA, Romero Y, Smyrk TC, Talley NJ. Swallowed fluticasone improves histologic but not symptomatic response of adults with eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):742-749.e1. doi: 10.1016/j.cgh.2012.03.018. Epub 2012 Apr 1. PMID 22475741
- [Background] Asher Wolf W, Dellon ES. Eosinophilic esophagitis and proton pump inhibitors: controversies and implications for clinical practice. Gastroenterol Hepatol (N Y). 2014 Jul;10(7):427-32. PMID 25904830
- [Background] Moawad FJ, Veerappan GR, Dias JA, Baker TP, Maydonovitch CL, Wong RK. Randomized controlled trial comparing aerosolized swallowed fluticasone to esomeprazole for esophageal eosinophilia. Am J Gastroenterol. 2013 Mar;108(3):366-72. doi: 10.1038/ajg.2012.443. Epub 2013 Feb 12. PMID 23399553
- [Background] Bullock JZ, Villanueva JM, Blanchard C, Filipovich AH, Putnam PE, Collins MH, Risma KA, Akers RM, Kirby CL, Buckmeier BK, Assa'ad AH, Hogan SP, Rothenberg ME. Interplay of adaptive th2 immunity with eotaxin-3/c-C chemokine receptor 3 in eosinophilic esophagitis. J Pediatr Gastroenterol Nutr. 2007 Jul;45(1):22-31. doi: 10.1097/MPG.0b013e318043c097. PMID 17592361
- [Background] Blanchard C, Mingler MK, Vicario M, Abonia JP, Wu YY, Lu TX, Collins MH, Putnam PE, Wells SI, Rothenberg ME. IL-13 involvement in eosinophilic esophagitis: transcriptome analysis and reversibility with glucocorticoids. J Allergy Clin Immunol. 2007 Dec;120(6):1292-300. doi: 10.1016/j.jaci.2007.10.024. PMID 18073124
- [Background] Park JY, Zhang X, Nguyen N, Souza RF, Spechler SJ, Cheng E. Proton pump inhibitors decrease eotaxin-3 expression in the proximal esophagus of children with esophageal eosinophilia. PLoS One. 2014 Jul 2;9(7):e101391. doi: 10.1371/journal.pone.0101391. eCollection 2014. PMID 24988451
- [Background] Zhang X, Huo X, Yu C, Zhang Q, Nadatani Y, Tamagawa Y, et al. Omeprazole and fluticasone inhibit IL-13-stimulated eotaxin-3 expression by esophageal epithelial cells through different mechanisms and with additive effects: Rationale for combining PPIs with topical steroids for EoE patients. Gastroenterology 2015;148(4, Supplement 1):S-51.
- [Background] Dellon ES, Gonsalves N, Hirano I, Furuta GT, Liacouras CA, Katzka DA; American College of Gastroenterology. ACG clinical guideline: Evidenced based approach to the diagnosis and management of esophageal eosinophilia and eosinophilic esophagitis (EoE). Am J Gastroenterol. 2013 May;108(5):679-92; quiz 693. doi: 10.1038/ajg.2013.71. Epub 2013 Apr 9. PMID 23567357
- [Background] Papadopoulou A, Koletzko S, Heuschkel R, Dias JA, Allen KJ, Murch SH, Chong S, Gottrand F, Husby S, Lionetti P, Mearin ML, Ruemmele FM, Schappi MG, Staiano A, Wilschanski M, Vandenplas Y; ESPGHAN Eosinophilic Esophagitis Working Group and the Gastroenterology Committee. Management guidelines of eosinophilic esophagitis in childhood. J Pediatr Gastroenterol Nutr. 2014 Jan;58(1):107-18. doi: 10.1097/MPG.0b013e3182a80be1. PMID 24378521
- [Background] Dellon ES, Cotton CC, Gebhart JH, Higgins LL, Beitia R, Woosley JT, Shaheen NJ. Accuracy of the Eosinophilic Esophagitis Endoscopic Reference Score in Diagnosis and Determining Response to Treatment. Clin Gastroenterol Hepatol. 2016 Jan;14(1):31-9. doi: 10.1016/j.cgh.2015.08.040. Epub 2015 Sep 25. PMID 26404868
- [Background] Hirano I, Moy N, Heckman MG, Thomas CS, Gonsalves N, Achem SR. Endoscopic assessment of the oesophageal features of eosinophilic oesophagitis: validation of a novel classification and grading system. Gut. 2013 Apr;62(4):489-95. doi: 10.1136/gutjnl-2011-301817. Epub 2012 May 22. PMID 22619364

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03781596/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03781596/ICF_001.pdf